CLINICAL TRIAL: NCT04116931
Title: A Randomized Controlled Trial on the Switch From Ticagrelor to Clopidogrel in Acute Coronary Syndrome Patients After Percutaneous Coronary Intervention--OPTImal Management of Antithrombotic Agents: OPTIMA-5
Brief Title: OPTImal Management of Antithrombotic Agents: OPTIMA-5
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, Dr., MD, Ph.D, Director of CCU Ward, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 011
Record Dates: First submitted 2019-09-26; First posted 2019-10-07 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Acute Coronary Syndrome (ACS)
Keywords: Dual antiplatelet therapy (DAPT); Platelet function; Clopidogrel; Ticagrelor; Switch
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- clopidogrel-600 mg-12h (Experimental): clopidogrel 600 mg loading dose (LD) 12 hours after the last maintenance dose（MD） of ticagrelor followed by 75 mg MD daily
  Interventions: Drug: Switch ticagrelor to clopidogrel
- clopidogrel-600 mg-24h (Experimental): clopidogrel 600 mg loading dose (LD) 24 hours after the last maintenance dose（MD） of ticagrelor followed by 75 mg MD daily
  Interventions: Drug: Switch ticagrelor to clopidogrel
- clopidogrel-75 mg-12h (Experimental): clopidogrel 75 mg maintenance dose(MD) 12 hours after the last MD of ticagrelor
  Interventions: Drug: Switch ticagrelor to clopidogrel
- clopidogrel-75 mg-24h (Experimental): clopidogrel 75 mg maintenance dose（MD) 24 hours after the last MD of ticagrelor
  Interventions: Drug: Switch ticagrelor to clopidogrel

INTERVENTIONS:
Drug: Switch ticagrelor to clopidogrel — Switch ticagrelor to clopidogrel with 600 mg loading dose (LD)/75 mg maintenance dose（MD）12/24 hours after the last MD of ticagrelor
  Other Names: switch

SUMMARY:
This is a prospective, randomized, open-label clinical trial which will enroll 80 acute coronary syndrome (ACS) patients after Percutaneous Transluminal Coronary Intervention (PCI) in China. Patients on maintenance dosing (MD) of aspirin (100 mg/d) and ticagrelor (90 mg twice daily) will be divided into two groups switching from ongoing ticagrelor to clopidogrel 600 mg loading dose (LD)/ 75 mg MD according to their bleeding risk. Then each group will randomly switch at different times(24 hours/ 12 hours after the last MD of ticagrelor). Pharmacodynamic assessments are performed at baseline, and at 4h, 8h, 24h, 48h, 72h hours with platelet aggregation rate by Light Transmittance Aggregometry method (LTA). All patients are followed-up for 30 days.

DETAILED DESCRIPTION:
The primary endpoint of the study was platelet inhibition measured by Light Transmittance Aggregometry method(LTA). Secondary clinical endpoints included a 30-day major adverse cardiovascular endpoint (MACE) defined as a composite of cardiovascular death, recurrent myocardial infarction, target vessel revascularisation or stroke and individual components of the MACE. Safety endpoints of 30-day TIMI major and minor bleed were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years.
* ACS patients.
* Patients who are treated with ticagrelor and do not tolerate it.
* Volunteer to participate and sign informed consent.
* Approved by national regulatory authorities ethics committees.

Exclusion Criteria:

* Patients who are contraindicated, intolerant or resistant to clopidogrel.
* History of hematological disease or bleeding tendency; platelet count < 100 × 10^9 cells/L, or > 600 × 10^9 cells/L, hemoglobin < 100 g/L.
* Abnormal liver or kidney function (ALT > 3 ULN; estimated CrCl < 30 ml/min calculated by Cockcroft-Gault equation); diagnosed severe pulmonary disease.
* Patients in need of drugs which affect the efficacy of clopidogrel such as miconazole, ketoconazole, andfluconazole.
* Malignancies or other comorbid conditions with life expectancy less than 1 year.
* Pregnant or lactating woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of platelet aggregation between different time points | baseline,4 hours,8 hours,24 hours,48 hours,72 hours
  Regional differences between blood samples from each subjects of different groups by LTA.The results of LTA are reported in platelet aggregation rate(%).Platelet aggregation was induced by0.5mg/ml arachidonic acid (AA).

SECONDARY OUTCOMES:
Rate of clinical endpoint event | 30 days
  Secondary clinical endpoints included a 30-day major adverse cardiovascular endpoint (MACE) defined as a composite of cardiovascular death, recurrent myocardial infarction, target vessel revascularisation or stroke and individual components of the MACE. Safety endpoints of 30-day TIMI major and minor bleed were also evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Chunjian Li, Dr, PhD, Principal Investigator — Principal Investigator
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No